CLINICAL TRIAL: NCT02282995
Title: Effect of Genetic Association With Functional Dyspepsia and Mood Disorders
Acronym: FDFDR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Justin Che-Yuen Wu, Professor, Chinese University of Hong Kong
Other Study IDs: FDFDR
Record Dates: First submitted 2014-04-17; First posted 2014-11-05 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Dyspepsia
Keywords: Functional dyspepsia; symptom response
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nine ml of blood will be used for the detection of biomarkers for functional dyspepsia through single nucleotide polymorphism (SNPs). The genotyping DNA will be isolated from whole blood samples by (FlexGene DNA kit, Qiagen). High-throughput genotyping will be performed on the serotonin 3A receptor polymorphism (rs1062613) and ghrelin CLOCK 3111C polymorphism (rs1801260). It will be analyzed by Applied Biosystems (ABI) 3730xl DNA Analyzer.
  Six ml of blood will be used for detection of plasma ghrelin and serotonin expression by ELISA.
  The remaining blood samples will be stored in the Laboratory of Institute of Digestive Diseases for tests stated in the Aim section, also for future studies for emerging diseases related to FGID.

GROUPS / COHORTS (4):
- •FDR-Relatives of FD patients: Relatives of FD patients. Patients may bring at most two FDRs to participate in this study.
  * Up to 20 ml of fasting blood sample will be collected
  * Serology test of Hp status will be performed for healthy volunteers and all FDRs
- •FDC-Healthy control: Healthy control. Controls who are self-referred to this study will be recruited.
  * Up to 20 ml of fasting blood sample will be collected
  * Fasting glucose test will be performed for FD patients
  * Serology test of Hp status will be performed for healthy volunteers and all FDRs
- •FD-Patients with FD: Patients with FD. Patients referred for OGD in Endoscopy Center, Prince of Wales Hospital, with symptoms suggestive of FGID will be invited to participate in this study.
  * Up to 20 ml of fasting blood sample will be collected
  * Fasting glucose test will be performed for FD patients
- •FDCR-Relatives of healthy controls: Relatives of healthy controls. Each participating control is required to bring at least one and up to two FDRs to participate in this study.
  * Up to 20 ml of fasting blood sample will be collected
  * Serology test of Hp status will be performed for healthy volunteers and all FDRs

SUMMARY:
Background:

Functional dyspepsia (FD) is one of the commonest digestive disorders. The pathophysiology of functional dyspepsia is uncertain. Risk factors include genetics, gender, age, helicobacter pylori infection, etc. However, few reported the association of genetic contribution to the development of FD and mood disorder.

Indication:

Functional dyspepsia patients

Study center(s):

Prince of Wales Hospital, Hong Kong

Aims:

* To evaluate genetic factors on development of functional dyspepsia & common mood disorders
* To evaluate genetic factors on the severity of function dyspepsia & mood disorders
* To develop a diagnostic test for classification of functional dyspepsia by plasma ghrelin and serotonin expression
* To collect sleep data for future use
* To save blood sample for future retrospective diagnostic or genetic examination

Study design:

Case-control cross sectional study

Number of subjects:

Total of 1200 subjects (300 FD patients + 300 relatives of FD patients FDR) and (300 Controls + 300 FDR)

Patient population:

Functional dyspepsia patients age 18-60

Duration of study:

1 May 2012 - 30 April 2013

Primary variable(s):

Genetic polymorphisms of targeted genes, plasma ghrelin and serotonin expression

Secondary variable(s):

FD global symptom assessment and symptom scores

Number of visits: 1

Hypotheses:

* Shared genetic factors contribute to the development of FD and common psychological disorders
* FD patients contribute to suppression of plasma ghrelin and serotonin expression compared to healthy controls

DETAILED DESCRIPTION:
Methods:

All subjects will participate in (1) Demographic assessment, (2) Questionnaires administration and (3) Blood sample collection. The three steps must be completed within 2 weeks.

1. Demographic assessment

   * Demographic: age, gender
   * Anthropometric measurements: body mass index, height, weight
   * Smoke and drink habit
   * Comorbidity and medical history
2. Questionnaires administration

   * A combined functional gastrointestinal (GI) symptom questionnaire (FGISQ) based on recall of the past 7 days will be used for assessment all GI symptoms including regurgitation, heartburn, epigastric pain, postprandial fullness, abdominal pain, diarrhea, constipation etc. All questions use a 4-point (0-3) Likert scale.
   * FGI Screening Questionnaire (v.3, 20101011) for screening of functional gastrointestinal disorder according to Rome III criteria. The questionnaire incorporate a GERD diagnostic questionnaire GERDQ (Chinese version)
   * Hospital Anxiety and Depression Scale (HADS) for a self administered scale for seven covering depression and seven covering anxiety.
   * Psychological disorder: Patient Health Questionnaire (PHQ) will be used for screening of concomitant psychological disorder such as depression and generalized anxiety disorder.
   * The Epworth Sleepiness Scale, Pittsburgh sleep quality index, and General Sleep Quality Questionnaire to collect sleep data for future use.
3. Blood sample collection

   * Up to 20 ml of fasting blood sample will be collected for study aims 1-4.
   * Fasting glucose test will be performed for FD patients
   * Serology test of Hp status will be performed for healthy volunteers and all FDRs

Subjects who had fasting glucose test or serology test performed within one year before study enrollment can be exempted from repeating the tests if they refuse to repeat the tests. In such cases, their previous test results will be recorded and used in this study.

If the subjects are found to be positive as a result of Helicobacter pylori (Hp) serology test, a referral letter with prescription suggestion will be given to the subjects to seek proper medical care in the primary care setting. In current practice, Hp eradication is not mandatory for asymptomatic subjects.

Laboratory work:

Nine ml of blood will be used for the detection of biomarkers for functional dyspepsia through single nucleotide polymorphism (SNPs). The genotyping DNA will be isolated from whole blood samples by (FlexGene DNA kit, Qiagen). High-throughput genotyping will be performed on the serotonin 3A receptor polymorphism (rs1062613) and ghrelin CLOCK 3111C polymorphism (rs1801260). It will be analyzed by Applied Biosystems (ABI) 3730xl DNA Analyzer.

Six ml of blood will be used for detection of plasma ghrelin and serotonin expression for development of diagnostic test in classification of functional dyspepsia by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* All subject

  * Age 18-60
  * Provision of written consent

Additional to FD patient

* Symptoms fulfilling Rome III criteria of functional dyspepsia
* Negative upper endoscopy (oesophagogastroduodenoscopy or OGD) finding

Exclusion Criteria:

* All subject

  * History of cancer
  * Diabetes mellitus
  * History of gastric surgery
  * Acid suppressants or medications that affect motility in past 4 weeks
  * Organic disease as cause of dyspepsia (for subjects with dyspeptic symptom)

Additional to healthy volunteer

• Any gastrointestinal symptoms (including acid regurgitation, heartburn, epigastric pain, bloating sensation, constipation, abdominal pain, diarrhea) in the past 4 weeks

Additional to FD patient

* Frequent (once or more per week) acid reflux or heartburn symptoms
* Helicobacter pylori (Hp) infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients referred for OGD in Endoscopy Center, Prince of Wales Hospital, with symptoms suggestive of FGID or who participated in PI's previous clinical trials will be invited to participate in this study as FD patients.
  Patients not suffering from FGID will be identified from the gastrointestinal specialty clinic or Endoscopy Center, Prince of Wales Hospital as healthy volunteers. These patients may include those referred for GI malignancy screening.
  Study advertisement will be posted in public area of Prince of Wales Hospital, and on the educational website (www.digestion.hk) which is maintained by PI. Controls who are self-referred to this study will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2012-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Differences of genetic polymorphism in targeted genes in patients with FD and mood disorders | up to 48 months
  Differences of genetic polymorphism in targeted genes in patients with FD and mood

SECONDARY OUTCOMES:
Diagnosis of psychiatric disorder with PHQ and HADS | up to 48 months
  Diagnosis of psychiatric disorder with PHQ and HADS
Differences of plasma ghrelin and serotonin expression in FD patients and study controls. | up to 48 months
  Differences of plasma ghrelin and serotonin expression in FD patients and study controls.
Symptom scores | up to 48 months
  Symptom scores

CONTACTS AND LOCATIONS:
Overall Officials: Justin C.Y. Wu, MBChB(CUHK), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Chinese University of Hong Kong — http://www.cuhk.edu.hk